CLINICAL TRIAL: NCT00672334
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Study of the Effect of Sodium Bicarbonate on Postoperative Renal Function in Patients Undergoing Elective Cardiopulmonary Bypass
Brief Title: Sodium Bicarbonate in Cardiac Surgery Study
Acronym: Bic-MC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Rinaldo Bellomo, Director of ICU research, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT 2007-002223-32
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
Keywords: Cardiac surgery; Cardiopulmonary bypass; Oxidative stress; Acute renal dysfunction; Sodium bicarbonate
MeSH Terms: interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): sodium chloride at 0.5 mmol/kg loading pre-induction and then at 0.2 mmol/kg/hr over 24 hours after induction until the next day
  Interventions: Drug: Sodium Chloride
- 1 (Experimental): The active intervention is loading (05. mmol/kg) pre-surgery and continuous infusion of bicarbonate at 0.2 mmol/kg/hr for 24 hours after induction
  Interventions: Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Sodium Bicarbonate — In all patients body weight adjusted dose of study medication will be achieved by infusion of sodium bicarbonate at a dose of 0.5 mmol/kg body weight (=bolus) diluted in 250 mL over 1 hour immediately after the induction of anesthesia, prior to the first surgical incision followed by continuous intravenous infusion of 0.2 mmol/kg/hr (=maintenance) diluted in 1000 mL 23 hours (total dose of 5 mmol/kg over 24 hours).
  Other Names: Hypertonic bicarbonate
  Arms: 1
Drug: Sodium Chloride — In all patients body weight adjusted dose of study medication will be achieved by infusion of sodium chloride at a dose of 0.5 mmol/kg body weight (=bolus) diluted in 250 mL over 1 hour immediately after the induction of anesthesia, prior to the first surgical incision followed by continuous intravenous infusion of 0.2 mmol/kg/hr (=maintenance) diluted in 1000 mL 23 hours (total dose of 5 mmol/kg over 24 hours).
  Other Names: hyeprtonic sodium chloride
  Arms: 2

SUMMARY:
With over one million operations a year, cardiac surgery with cardiopulmonary bypass is one of the most common major surgical procedures worldwide (1). Acute kidney injury is a common and serious postoperative complication of cardiopulmonary bypass and may affect 25% to 50% of patients (2-4). Acute kidney injury carries significant costs (4) and is independently associated with increased morbidity and mortality (2,3). Even minimal increments in plasma creatinine are associated with an increase in mortality (5,6).

Multiple causes of cardiopulmonary bypass-associated acute kidney injury have been proposed, including ischemia-reperfusion, generation of reactive oxygen species, hemolysis and activation of inflammatory pathways (7-10). COMT LL genotype appears to increase the risk of vasodilatory shock and AKI after cardiac surgery. To date, no simple, safe and effective intervention to prevent cardiopulmonary bypass-associated acute kidney injury in a broad patient population has been found (11-14).

Urinary acidity may enhance the generation and toxicity of reactive oxygen species induced by cardiopulmonary bypass (10,15). Activation of complement during cardiac surgery (16) may also participate in kidney injury. Urinary alkalinization may protect from kidney injury induced by oxidant substances, iron-mediated free radical pathways, complement activation and tubular hemoglobin cast formation (9,17,18). Of note, increasing urinary pH - in combination with N-acetylcysteine (19,20) or without (21) - has recently been reported to attenuate acute kidney injury in patients undergoing contrast-media infusion.

In a pilot double-blind, randomized controlled trial the investigators found sodium bicarbonate to be efficacious, safe, inexpensive and easy to administer. These findings now need to be confirmed or refuted by further clinical investigations in other geographic and institutional settings.

Accordingly, the investigators hypothesized that urinary alkalinization might protect kidney function in patients at increased risk of acute kidney injury undergoing cardiopulmonary bypass needs to be confirmed in an international multicenter, double-blind, randomized controlled trial of intravenous sodium bicarbonate.

DETAILED DESCRIPTION:
Renal impairment following cardiopulmonary bypass is common. While most of these patients do not require either short or long term renal replacement, the mortality of patients with acute renal failure is substantially greater than those who do not develop renal dysfunction.

In a pilot double-blind, randomized controlled trial we found sodium bicarbonate to be efficacious, safe, inexpensive and easy to administer. These findings now need to be confirmed or refuted by further clinical investigations in other geographic and institutional settings.

There is evidence that sodium bicarbonate affects the cardiovascular, respiratory and immune systems and may be of benefit to patients undergoing cardiac surgery.

Study Design - overview and rationale Patients will be randomised to receive sodium bicarbonate from the induction of anaesthesia until 24 hours postoperatively, or a placebo (sodium chloride).

Serum creatinine is the most commonly used clinical indicator of renal function along with urine output. Both will be measured for several days postoperatively - the time period during which renal impairment is most likely to develop.

Randomisation The randomisation will be based on random numbers generated by computer. Once consent is obtained, the allocation of either treatment with sodium bicarbonate or placebo will be organised by an independent person (clinical trials pharmacist) who will dispense the coded and blinded infusion bags (shrink-wrapped in extra black plastic bags). This will be delivered to the anaesthetic staff looking after the patient in theatre, and the ICU nurse caring for the patient postoperatively.

20 ml samples of heparinised blood and urine will be taken from the arterial line or urine catheter. Samples will be taken immediately after the preoperative insertion of the arterial/urine catheter, at 6, 24, 48, 72, 96 and 120 hours after commencement of cardiopulmonary bypass. Immediately following collection, the preoperative, 6 and 24 hour blood and urine will be centrifuged at low speed to separate the plasma from the cellular components. Urine and plasma and full-blood (for COMT polymorphism) will be stored in aliquots (where necessary) at -70 degrees prior to batch analysis.

The following variables will be obtained:

Code for patient, gender and age. Date and time of admission to ICU Operative procedure and date and time on and off cardiopulmonary bypass Preoperative assessment of left ventricular function, Comorbidities, Pre-, intra- and post-operative medication, Markers of renal function and COMT polymorphism as described above, Doses of frusemide administered (or rate of frusemide infusion) Use of inotropes or vasopressors Cardiac output whenever measured for clinical purposes in the first 24 hours postoperatively Requirement of renal replacement therapy Urine output in each 6 hour period during the presence of urine catheter Acid base status and electrolytes at baseline, 6 and 24 hours after commencement of cardiopulmonary bypass, Time of intubation and extubation, Date and time of arrival on and discharge from ICU and hospital, death Resources required The principle of the study has been discussed with the involved cardiac anaesthetists, cardiac surgeons, intensivists and intensive care nurses, who have offered their co-operation. ICU research nurse to allocate patients and collect clinical data. Pharmacy will be required to prepare drug and placebo infusion bags. Clinical pathology will be required to perform 24 hour creatinine clearance estimation (in addition to those tests clinically indicated) Protocol violations All protocol violations will be recorded. It will then be decided whether the nature of such violation had been such that the patient should be excluded from primary data analysis. Such evaluation will be blinded to treatment.

Withdrawal The treating clinician will have the right to withdraw the patient from the study if he or she believes that continued participation is jeopardising the patient's well being.

Ethical Issues sodium bicarbonate used in this study is considered to be very safe as has been demonstrated by its widespread clinical use in the management of critically ill patients with metabolic acidosis. We consider the potential benefit of this treatment theoretically significant. Given the balance of benefits and risks, we consider it ethical to proceed and seek informed consent.

Indemnity This is an investigator-initiated study and, accordingly, no commercial sponsor's indemnity has been provided.

Informed consent will be obtained from the patient prior to the operation by one of the investigators or the ICU research nurse. The clinical care of a patient who does not consent for any reason will not be affected.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgical patients in whom the use of cardiopulmonary bypass was planned and:
* Written informed consent of patient
* Age >18 years
* And having at least one ore more of the following risk factors for postoperative AKI:

  * Age =/>70 years
  * Preoperative plasma creatinine >120 µmol/L New York Heart Association class III / IV or LVEF <35%
  * Insulin dependent diabetes mellitus
  * Valve surgery (with or without coronary artery bypass graft)
  * Redo cardiac surgery

Exclusion Criteria:

* Cardiac surgical patients will not be considered eligible if:
* An emergency operation is indicated (within 24 hours after hospital admission or on intra-aortic balloon pump) or
* Pregnancy is confirmed or breastfeeding is present or
* A renal allograft is present or
* Preoperative acute renal failure within 6 weeks (acute rise in serum creatinine >50% from baseline) is present or
* Pre-operative end stage renal disease (serum creatinine >300 µmol/L) is present or
* Chronic moderate to high dose corticosteroid therapy (>10 mg/d prednisone or equivalent) is present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing an increase in serum creatinine > 25% or >44µmicromol/L from baseline to peak level after adjustment for relevant baseline characteristics | within first two-five postoperative days.

SECONDARY OUTCOMES:
Proportion of patients developing an increase in serum creatinine greater than 50% from baseline to peak level after adjustment for relevant baseline characteristics | within first two-five postoperative days
Proportion of patients developing an increase in serum creatinine greater than 100% from baseline to peak level after adjustment for relevant baseline characteristics | within first two-five postoperative days
Change in serum creatinine from baseline to peak level after adjustment for relevant baseline characteristics | within first two-five postoperative days
Proportion of patients developing any of the RIFLE criteria: R, I or F after adjustment for relevant baseline characteristics | within first five postoperative days
Proportion of patients developing any of the AKI stages: 1, 2 or 3 (using network definition)after adjustment for relevant baseline characteristics | within 48 hours postoperatively
Change in serum urea from baseline to peak | within first two-five postoperative days
Change in NGAL from baseline to peak | within first 24 postoperatively
Change in electrolyte status from baseline to peak | within first 24-48hrs postoperatively
Requirement of renal replacement therapy | within first postoperative days
Length of ventilation | from commencement to end of intubation
Length of stay in Intensive care | from admission to discharge from Intensive care
Length of stay in hospital | from admission to discharge from hospital
Hospital-Mortality | during hospital stay
90-day mortality | during 90 days postoperatively
COMT polymorphism | sampling at induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MD, FRACP, Study Chair — Austin Health, Melbourne, Australia; Michael Haase, MD, Principal Investigator — Charité-University Medicine (Berlin, Germany); Sean M Bagshaw, MD, Principal Investigator — University of Alberta, Edmonton, Canada; Patrick Murray, MD, Principal Investigator — University Clinic Dublin, Dublin, Ireland
Locations (4):
- Austin Health, Melbourne, Victoria, Australia
- University of Alberta, Edmonton, Alberta, Canada
- Charité University Medicine, Berlin, State of Berlin, Germany
- University Clinic Dublin, School of Medicine and Medical Science, Dublin, Dublin, Ireland

REFERENCES:
- [Derived] Elitok S, Kuppe H, Devarajan P, Bellomo R, Isermann B, Westphal S, Kube J, Albert C, Ernst M, Kropf S, Haase-Fielitz A, Haase M. Urinary Neutrophil Gelatinase-Associated Lipocalin/Hepcidin-25 Ratio for Early Identification of Patients at Risk for Renal Replacement Therapy After Cardiac Surgery: A Substudy of the BICARBONATE Trial. Anesth Analg. 2021 Dec 1;133(6):1510-1519. doi: 10.1213/ANE.0000000000005741. PMID 34543256
- [Derived] Elitok S, Devarajan P, Bellomo R, Isermann B, Haase M, Haase-Fielitz A. NGAL/hepcidin-25 ratio and AKI subtypes in patients following cardiac surgery: a prospective observational study. J Nephrol. 2022 Mar;35(2):597-605. doi: 10.1007/s40620-021-01063-5. Epub 2021 May 24. PMID 34028701
- [Derived] Haase M, Haase-Fielitz A, Plass M, Kuppe H, Hetzer R, Hannon C, Murray PT, Bailey MJ, Bellomo R, Bagshaw SM. Prophylactic perioperative sodium bicarbonate to prevent acute kidney injury following open heart surgery: a multicenter double-blinded randomized controlled trial. PLoS Med. 2013;10(4):e1001426. doi: 10.1371/journal.pmed.1001426. Epub 2013 Apr 16. PMID 23610561
- [Derived] Haase-Fielitz A, Plass M, Kuppe H, Hetzer R, Ostland V, Westphal S, Hoffmann J, Prowle J, Mertens PR, Westerman M, Bellomo R, Haase M. Low preoperative hepcidin concentration as a risk factor for mortality after cardiac surgery: a pilot study. J Thorac Cardiovasc Surg. 2013 May;145(5):1380-6. doi: 10.1016/j.jtcvs.2012.09.003. Epub 2012 Oct 9. PMID 23062413
- [Derived] Haase-Fielitz A, Mertens PR, Plass M, Kuppe H, Hetzer R, Westerman M, Ostland V, Prowle JR, Bellomo R, Haase M. Urine hepcidin has additive value in ruling out cardiopulmonary bypass-associated acute kidney injury: an observational cohort study. Crit Care. 2011 Aug 4;15(4):R186. doi: 10.1186/cc10339. PMID 21816077